CLINICAL TRIAL: NCT04887376
Title: Additive Effect of Mirror Therapy on Effects of Cross-Education of Muscle Strength of Neuromuscular Electrical Stimulation In Hemiplegic Patients
Brief Title: Mirror Therapy and Cross-Education of Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstPMRTRH-MT
Record Dates: First submitted 2021-05-07; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Cerebrovascular Stroke; Muscle Weakness
Keywords: Cross-education; Neuromuscular electrical stimulation; Mirror Therapy
MeSH Terms: conditions — Stroke; Muscle Weakness

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy (Active Comparator): Participants were asked to sit with their knee joints in full extension and both ankle joints in a neutral position. Five sessions of neuromuscular electrical stimulation (NMES) were applied to the non-affected side ankle dorsiflexors. In addition to this application, mirror therapy was applied simultaneously with NMES.
  Interventions: Device: Mirror frame
- Control (Placebo Comparator): Participants were asked to sit with their knee joints in full extension and both ankle joints in a neutral position. Five sessions of neuromuscular electrical stimulation (NMES) were applied to the non-affected side ankle dorsiflexors.
  Interventions: Device: Control

INTERVENTIONS:
Device: Mirror frame — Combined Mirror and NMES therapy
  Arms: Mirror Therapy
Device: Control — Only NMES therapy
  Arms: Control

SUMMARY:
This study was conducted to determine whether mirror therapy has an additive effect on cross-education of the strength of neuromuscular electrical stimulation (NMES) in patients with hemiplegia. As an outcome measure, the ankle dorsiflexion strength of hemiplegic patients was measured.

DETAILED DESCRIPTION:
A total of 29 patients, 7 women, and 22 men were included according to the inclusion and exclusion criteria. The patients were randomly assigned to the control group (n = 14) and the Mirror group (n = 15). Five sessions of neuromuscular electrical stimulation, unaffected side ankle dorsiflexors were applied to the patients in both groups. In addition to the NMES, mirror therapy was applied to the experimental group simultaneously with NMES. Before and after treatment, both ankle dorsiflexor strength was measured with a force sensor. For force measurements, a force transducer (FC2211-0000-0100-L Compression Load Cell, TE Connectivity company, France) was used. Force transducer signals were received with a data acquisition device (POWERLAB® data acquisition system ADInstruments, Oxford, UK) and evaluated offline on the computer. The measurement values were expressed in kilogram.force (kg.f) and this value was normalized according to body weight.

ELIGIBILITY:
Inclusion Criteria:

* Cases with stroke duration ≥ 1 month
* Ability to walk at least 10m (functional ambulation scale ≥3)
* Age range 18-75 years
* Hemorrhagic or ischemic stroke
* Brunnstrom stage ≥4 for lower limb
* Unilateral stroke
* Cooperating with the examination and tests

Exclusion Criteria:

* Mini Mental State Assessment score <21
* Severe spasticity (MAS = 4) in ankle dorsiflexors
* Have a contracture on ankle joint
* The presence of skin lesions in the application area
* Painful pathologies in the lower extremities
* Having visual field defects
* Active inflammatory, rheumatological or infectious disease
* Parent rhythm / conduction block problem in the heart
* Uncontrollable hypertension (Maxima> 140, Minima> 90)
* Presence of lower extremity fracture
* Peripheral nerve lesions such as polyneuropathy, radiculopathy
* Finding or suspected active deep vein thrombosis
* History of deep vein thrombosis and pulmonary embolism

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change of ankle dorsiflexor isometric muscle strength | Change from Baseline muscle strength at 6 days
  Force transducer used for measuring maximum voluntary ankle dorsiflexion force. The force unit is kilogram.force

SECONDARY OUTCOMES:
Change of Lower Extremity Brunnstrom score | Change from Baseline Brunnstrom score at 6 days
  It evaluates the developmental stages of synergy patterns, muscle tone and isolated movements of the patients in the lower extremities. Patients are categorized between Stage-1 and 6. Stage 1: Flaccidity; Stage 6: Spasticity Disappears and Coordination Reappears
Change of Modified Ashworth Scale score | Change from Baseline Modified Ashworth Scale score at 6 days
  Modified Ashworth Scale was used for assessment spasticity. Modified Ashworth Scale scores are varied between 0 and 4: 0 points, no increase in muscle tone; 4 points indicate spasticity with a degree of rigidity.
Change of Functional Ambulation Scale score | Change from Baseline Functional Ambulation Scale score at 6 days
  The Functional Ambulation Classification (FAC) is a method for classifying mobility. The FAC has six categories ranging from 0 (non-functional ambulation) to 5 (independent).
Change of Timed Up and Go Test score | Change from Baseline Timed Up and Go Test score at 6 days
  It is a test that evaluates the patient's static and dynamic balance, mobility and walking ability. The test's score is the time in seconds it takes the subject takes to complete the test.

CONTACTS AND LOCATIONS:
Overall Officials: Ilhan Karacan, Assoc Prof, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training & Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howatson G, Zult T, Farthing JP, Zijdewind I, Hortobagyi T. Mirror training to augment cross-education during resistance training: a hypothesis. Front Hum Neurosci. 2013 Jul 24;7:396. doi: 10.3389/fnhum.2013.00396. eCollection 2013. PMID 23898251
- [Background] Zult T, Goodall S, Thomas K, Solnik S, Hortobagyi T, Howatson G. Mirror Training Augments the Cross-education of Strength and Affects Inhibitory Paths. Med Sci Sports Exerc. 2016 Jun;48(6):1001-13. doi: 10.1249/MSS.0000000000000871. PMID 26765630
- [Background] Sariyildiz M, Karacan I, Rezvani A, Ergin O, Cidem M. Cross-education of muscle strength: cross-training effects are not confined to untrained contralateral homologous muscle. Scand J Med Sci Sports. 2011 Dec;21(6):e359-64. doi: 10.1111/j.1600-0838.2011.01311.x. Epub 2011 Apr 18. PMID 21496110
- [Background] Lee D, Lee G. Effect of afferent electrical stimulation with mirror therapy on motor function, balance, and gait in chronic stroke survivors: a randomized controlled trial. Eur J Phys Rehabil Med. 2019 Aug;55(4):442-449. doi: 10.23736/S1973-9087.19.05334-6. Epub 2019 Mar 22. PMID 30916531
- [Background] Kim H, Lee G, Song C. Effect of functional electrical stimulation with mirror therapy on upper extremity motor function in poststroke patients. J Stroke Cerebrovasc Dis. 2014 Apr;23(4):655-61. doi: 10.1016/j.jstrokecerebrovasdis.2013.06.017. Epub 2013 Jul 16. PMID 23867040
- [Background] Ji SG, Cha HG, Kim MK, Lee CR. The effect of mirror therapy integrating functional electrical stimulation on the gait of stroke patients. J Phys Ther Sci. 2014 Apr;26(4):497-9. doi: 10.1589/jpts.26.497. Epub 2014 Apr 23. PMID 24764619